CLINICAL TRIAL: NCT02788370
Title: Cardiopulmonary Response to Conical Positive Expiratory Breathing During Exercise in Older People.
Brief Title: Cardiopulmonary Response to Conical-PEP Breathing During Exercise in Older People.
Acronym: CPEPolder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Chatchai Phimphasak, School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PHD/0082/2556.1
Record Dates: First submitted 2016-05-26; First posted 2016-06-02 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Aging
Keywords: Positive expiratory pressure; Cardiopulmonary responses; Exercise; Older people
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham-PEP breathing (Sham Comparator): Patients will perform a constant work load cycling test with sham-positive expiratory pressure breathing util symptom limit.
  Interventions: Other: Constant work load cycling test
- Conical-PEP breathing (Experimental): Patients will perform a constant work load cycling test with positive expiratory pressure breathing using a conical positive expiratory pressure device until symptom limit.
  Interventions: Device: a conical positive expiratory pressure device; Other: Constant work load cycling test

INTERVENTIONS:
Device: a conical positive expiratory pressure device — The CPEP device will be connected to respiratory transducer for generating positive expiratory pressure with therapeutic rang (5 to 20 cm H2O).
  Other Names: CPEP deice
  Arms: Conical-PEP breathing
Other: Constant work load cycling test — Participants will per form constant work load cycling test until symptom limit with 50 to 60 rpm. The termination criteria include
  1. sever breathlessness (>5 /10 score of modified Borg scale)
  2. leg fatigue (can not maintain speed between 50 to 60 rpm)
  3. Hear rate (HR) >80 % age-predicted maximum HR
  4. Exercise time up to 10 minutes
  5. Other symptom that stated by American thoracic Society(2002)

SUMMARY:
Aim of this study is to compare cardiopulmonary response to conical-PEP breathing during exercise in older people.

DETAILED DESCRIPTION:
It is known that all most structures and physiological functions deteriorate with age, leading to decrease exercise performance, functional decline and gradual decrease of physical activity in aging.

The most essential change of respiratory physiology are: dilatation of alveoli, enlargement of air space, decrease gas exchange surface area, loss of supporting tissue for distal airway (senile emphysema), decrees of chest wall compliance and decrease of respiratory muscle strength. These changes leading to decrease lung elastic recoil, increase residual volume and functional capacity, and increase work of breathing at rest. In addition, such changes affect respiratory function, especially dynamic hyperinflation (DH) development which could be one of the factors relate to dyspnea during exercise in aging Positive expiratory pressure (PEP) therapy for DH treatment during exercise was reported in several studies.

It is possible that PEP breathing may improve cardiopulmonary response to exercise in older people.

ELIGIBILITY:
Inclusion Criteria:

* Elder age between 60 to 80 years old with normal spirometry

Exclusion Criteria:

* They are diagnose with cardiovascular disease and, i.e. valvular heart disease, coronary heart disease, congenital heart disease, myocardial heart disease, uncontrolled hypertension, hyperlipidemia; or, present abnormal sign of heart problems previous month, such as chest pain, arrhythmia, abnormal ECG.
* They are impair balance from neuromuscular, musculoskeletal, or vestibular problem affecting cycling and walking.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of Inspiratory capacity (IC) | resting, immediate post exercise test and end recovery period of 10 minutes
  Participants will be measured IC with slow vital capacity maneuver following American thoracic Society (ATS) and European Respiratory Society (ERS) statement for spirometry (2005).

SECONDARY OUTCOMES:
Change of Slow vital capacity (SVC) | resting, immediate post exercise test and end recovery period of 10 minutes
  Participants will be measured SVC with slow vital capacity maneuver following American thoracic Society (ATS) and European Respiratory Society (ERS) statement for spirometry (2005).
Change of respiratory rate (RR) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The RR will be measured by a flow transducer of BioPAC system MP 36. The RR will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute
Change of hear rate (HR) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  Participants will be continuously recorded EKG by the BioPAC system MP 36 The HR will be collected from EKG. Moreover, real time EKG with HR will be measured by bedside monitor for termination criteria .
Change of inspiratory time (Ti) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The Ti will measure by a flow transducer of BioPAC system MP 36. The Ti will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute
Change of expiratory time (Te) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The Te will measure by a flow transducer of BioPAC system MP 36. The Te will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute
Change of inspiratory and expiratory time ratio (IE ratio) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The IE ratio will measure by a flow transducer of BioPAC system MP 36. The IE ratio will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute
Change of tidal volume (VT) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The VT will measure by a flow transducer of BioPAC system MP 36. The VT will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute
Change of expiratory minute ventilation (VE) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The VE will calculate from RR and VT and will present at resting, during exercise every minute, end exercise and every minute in recovery period for 10 minute
Change of mean expiratory flow rate (MEF) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The MEF will measure by a flow transducer of BioPAC system MP 36. The MEF will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute.
Change of peak expiratory flow rate (PEF) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The PEF will measure by a flow transducer of BioPAC system MP 36. The PEF will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute.
Change of mean expiratory pressure (MEP) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The MEP will measure by a pressure transducer of BioPAC system MP 36. The MEP will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute.
Change of peak expiratory pressure (PEP) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  The PEP will measure by a pressure transducer of BioPAC system MP 36. The PEP will continuously measure throughout resting, during exercise, end exercise and recovery period fro 10 minute.
Change of pule oxygen saturation (SpO2) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  Participants will be continuously measured SpO2 throughout the test. Researcher will collect SpO2 at resting, every minute during exercise, end exercise test and every minute of recovery period for 10 minutes.
Change of end tidal carbon dioxide pressure (PetCO2) | Resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  Participants will be continuously measured PetCO2 throughout the test. Researcher will collect PetCO2 at resting, every minute during exercise, end exercise test and every minute of recovery period for 10 minutes.
Change of rating perceive of breathlessness (RPB) | resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes
  Participant will rate RPB using a modified Borg dyspnea 10 scale at resting, during exercise every minute, end exercise test and every minute of recovery period for 10 minutes.
Change of leg fatigue | resting, , end exercise test and end recovery period
  Participant will rate their leg fatigue using a visual analog scale at resting, end exercise test and end recovery period for 10 minutes.
Change of systolic blood pressure (SBP) | resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes
  The SBP will be measured by a bedside monitor at resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes.
Change of diastolic blood pressure (DBP) | resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes
  The SBP will be measured by a bedside monitor at resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes.
Change of mean arterial pressure (MAP) | resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes
  The MAP will be measured by a bedside monitor at resting, immediate post exercise test and every 2 minutes during recovery period for 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Chulee U Jones, Ph.D., PT, Principal Investigator — School of Physical therapy, Faculty of Associated Medical Sciences, Khon Kaen University

IPD SHARING:
Plan to Share IPD: Undecided